CLINICAL TRIAL: NCT05134142
Title: Quality of Life and Function of Patients After Hemipelvectomy
Brief Title: Quality of Life and Function of Patients With Pelvic Tumors After Undergoing Hemipelvectomy
Status: Recruiting | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: PA12-1046; NCI-2021-11297 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); PA12-1046 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2021-11-11; First posted 2021-11-24 (Actual); Last update posted 2025-11-06 (Actual); Status verified 2025-11

CONDITIONS: Malignant Primary Pelvic Neoplasm
MeSH Terms: interventions — Exercise Test

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Observational (Physical tests, questionnaires, record review): Patients undergo physical performance assessments and complete quality of life assessments and questionnaires pre-hemipelvectomy, at 6 weeks post-hemipelvectomy, and then every 3 months up to 12 months and yearly thereafter for 10 years. Patients who are 1 year out from surgery complete pain-related questionnaires once. Patients who have already undergone hemipelvectomy prior to enrollment undergo medical record review.
  Interventions: Other: Electronic Health Record Review; Other: Physical Performance Testing; Other: Quality-of-Life Assessment; Other: Questionnaire Administration

INTERVENTIONS:
Other: Electronic Health Record Review — Undergo medical record review
Other: Physical Performance Testing — Undergo physical performance testing
  Other Names: Physical Fitness Testing; Physical Function Testing
Other: Quality-of-Life Assessment — Complete assessments
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Complete questionnaire

SUMMARY:
This study aims to determine the functional outcomes of patients who underwent internal hemipelvectomy with or without reconstruction or external hemipelvectomy for pelvic tumors. Learning about the outcomes of these patients may help researchers determine the long-term effects of different types of hemipelvectomy procedures and may help improve quality of life.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine functions of patients who underwent internal hemipelvectomy with or without reconstruction or have had an external hemipelvectomy.

SECONDARY OBJECTIVES:

I. To determine factors that influence the functional outcomes of these patients following surgery.

II. Assess sexual and urinary function in patients who have undergone internal or external hemipelvectomy.

III. Determine whether type of surgery influences long-term sexual and urinary function.

OUTLINE:

Patients undergo physical performance assessments and complete quality of life assessments and questionnaires pre-hemipelvectomy, at 6 weeks post-hemipelvectomy, and then every 3 months up to 12 months and yearly thereafter for 10 years. Patients who are 1 year out from surgery complete pain-related questionnaires once. Patients who have already undergone hemipelvectomy prior to enrollment undergo medical record review.

ELIGIBILITY:
Inclusion Criteria:

* Patients within the institution who have undergone or will undergo a hemipelvectomy

Exclusion Criteria:

- None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients within the institution who have undergone or will undergo a hemipelvectomy.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2013-03-27 (Actual); Primary Completion 2027-04-30 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Functions of patients who underwent internal hemipelvectomy with or without reconstruction or have had an external hemipelvectomy | Through study completion, average of 1 year
  All continuous variables including the scoring systems will be described as mean with standard deviation or median with range. Frequencies and percentages will be obtained for all categorical variables. Pediatric participants' data measures will be collected and analyzed separately from the adult populations.

CONTACTS AND LOCATIONS:
Overall Officials: Valerae O Lewis, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M D Anderson Cancer Center website — http://www.mdanderson.org